CLINICAL TRIAL: NCT04653168
Title: A Single Dose, Open-Label Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Subcutaneous Injections of LY3041658 in Healthy Participants
Brief Title: A Study of LY3041658 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17745; I7P-MC-DSAE (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-12-03; First posted 2020-12-04 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06-15

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY3041658 Low Dose (Experimental): LY3041658 administered by subcutaneous (SC) injection.
  Interventions: Drug: LY3041658
- LY3041658 High Dose (Experimental): LY3041658 administered by SC injection.
  Interventions: Drug: LY3041658

INTERVENTIONS:
Drug: LY3041658 — Administered SC

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3041658 in healthy participants. The study will measure how the body absorbs, breaks down and gets rid of LY3041658.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs, and ECG.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Have Body mass index (BMI) within the range 18.5 - 35.0 kilograms per square meter (kg/m2) (inclusive).

Exclusion Criteria:

* Have a significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, immune, neurological, dermatological, or psychiatric disorder capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the Study intervention or interfering with the interpretation of data.
* Have self-perceived dullness or loss of sensation on either side of their abdomen.
* Have any condition that could affect pain perception from an injection.
* Have excessive tattoos or scars over the abdomen, or other factors (eg, rash, excessive folds of skin) that, in the investigator's opinion, would interfere with injection site assessments.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants With incidence and severity of Injection Site Reaction (ISR) | Baseline up to Day 15
  Number of Participants With incidence and severity of ISR
Visual Analog Scale (VAS) Score for Injection Site Pain | Baseline up to Day 1
  VAS Score for Injection Site Pain

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3041658 | Predose up to day 85 postdose
  PK: Cmax of LY3041658
PK: Area Under the Concentration Versus Time Curve (AUC) from time 0 to infinity of LY3041658 | Predose up to day 85 postdose
  PK: AUC(0-inf) of LY3041658

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No